CLINICAL TRIAL: NCT02306044
Title: Bleeding Prediction in Thrombocytopenia Using Platelet Indices, Platelet Aggregometry and a Standardized Bleeding Questionnaire
Brief Title: Bleeding Prediction in Thrombocytopenia
Status: Completed | Type: Observational
Sponsor: Pernille Just Vinholt (Other)
Responsible Party: Sponsor-Investigator, Pernille Just Vinholt, MD, Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: s-20120088
Record Dates: First submitted 2014-11-24; First posted 2014-12-03 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Thrombocytopenia
Keywords: Bleeding; Platelet indices; Platelet aggregometry; Bleeding questionnaire
MeSH Terms: conditions — Thrombocytopenia; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to investigate whether platelet indices from automated haematology equipment, whole blood impedance aggregometry and a standardized bleeding questionnaire predict bleeding in admitted patients with thrombocytopenia of various causes.

DETAILED DESCRIPTION:
Thrombocytopenia is a risk factor for bleeding, but studies concerning markers for stratification of bleeding risk among thrombocytopenic patients are lacking. This prospective observational cohort study investigates risk factor for bleeding in admitted patients with thrombocytopenia of various causes.

ELIGIBILITY:
Inclusion Criteria:

* Admitted patients with thrombocytopenia
* Age ≥18 years
* Platelet count below 80 x109/L

Exclusion Criteria:

* Platelet transfusion within the previous 14 days,
* surgery or trauma within the previous 7 days
* Unable to give informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Admitted patients with thrombocytopenia of any cause
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Mean platelet volume | 30 days
  Mean platelet volume (femtolitre (fL))

SECONDARY OUTCOMES:
Platelet count | 30 days
  Platelet count ( x10'9/L)
immature platelet fraction | 30 days
  immature platelet fraction (%)
Bleeding questionnaire | 30 days
  Bleeding score based on the condensed MCMDM-1 VWD bleeding questionnaire
Platelet aggregation | 30 days
  Platelet aggregation by Multiplate Analyzer (aggregation units* min)

CONTACTS AND LOCATIONS:
Overall Officials: Pernille J Vinholt, MD, Principal Investigator — Odense University Hospital